CLINICAL TRIAL: NCT04459026
Title: Comparative Study Between Different Routes of Ropivacaïne Administration to Reduce Post-operative Pain in Gynecological Laparoscopy, a Double Blind Randomized Trial.
Brief Title: Comparison of Administation Routes of Ropivacaine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Prof Yves Jacquemyn, Professor Jacquemyn, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ropivacaine
Record Dates: First submitted 2018-02-28; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Postoperative Pain
Keywords: ropivacaine; laparoscopy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: We will be using ropivacaine - naropin 7,5mg/ml, a local anaesthetic of the amide type. The administered dose of this local anaesthetic will be 3mg/kg for each patient. Depending on the study group the patient belongs to, this dose will be given in full by either local injection at the trocar entry points or by intraperitoneal injection or it will be divided between both injection sites
Who Masked: Participant, Investigator
Masking Description: The participant won't know to what study group they are assigned and will be under general anaesthesia. The study medication will be prepared in the operating room right before use. This means that neither the anaesthesiologist nor the surgeon, performing the surgery, are blinded. The investigators filling in the questionnaires, the patients or the nurses of the recovery room will always be blinded to the study groups, as will the nurse contacting the patients for the follow up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group A - combination (Experimental): Group A patients will receive intra-abdominal instillation 0.75% Ropivacaine 2 mg / kg in 200 ml of NaCl through the trocars and 2) Infiltration of the surgical wounds at the trocar sites with 0.75% Ropivacaine 1 mg / kg in 20 ml of NaCl
  Interventions: Procedure: combination
- Group B - infiltration (Experimental): Group B patients will receive infiltration of the surgical wounds at the trocar sites with 0.75% Ropivacaine 3 mg / kg in 20 ml of NaCl.
  Interventions: Procedure: infiltration
- Group C - instillation (Active Comparator): Group C patients will receive intra-abdominal instillation 0.75% Ropivacaine 3 mg / kg in 200 ml of NaCl through the trocars.
  Interventions: Procedure: instillation

INTERVENTIONS:
Procedure: combination — instillation and infiltration of ropivacaine
  Other Names: ropivacaine intraperitoneal and local
  Arms: group A - combination
Procedure: infiltration — local infiltration ropivacaine
  Other Names: ropivacaine local
  Arms: Group B - infiltration
Procedure: instillation — intraperitoneal ropivacaine instillation
  Other Names: intraperitoneal ropivacaine
  Arms: Group C - instillation

SUMMARY:
The purpose of this study is to evaluate the effect of different routes of local anaesthesia administration in laparoscopic procedures to reduce post-operative pain (intra-peritoneal infusion of Ropivacaine 0.75%, port site injection of Ropivacaine 0.75% or a combination of both techniques), through a randomized one-center double-blinded study.

DETAILED DESCRIPTION:
Research Question What is the best route of Ropivacaine administration in laparoscopic procedures in decreasing post-operative pain? Is it port site injection, intra-peritoneal instillation of local anesthetics or is it a combination of both routes? Our hypothesis is that a combination of port site injection and intra-peritoneal instillation of local anesthetics will be more effective in lowering pain the first 24 hours after surgery.

3. Characteristics of the patient population Inclusion criteria

1. Elective gynecologic laparoscopy for benign conditions at Antwerp University Hospital.
2. Successful laparoscopy without surgical or anesthetic complications.
3. Female
4. 18-70 years
5. ASA( American Society of Anesthesia) I-II Exclusion criteria

(1) Hypersensitivity to anaesthetics of the amide-type (2) Obesity, BMI > 35 (3) Patients with chronic use of analgesics / chronic pain (4) Patients with an abnormal liver function (5) Urgent surgical procedures (6) Pregnancy (this means we only include patients who use contraceptives, are sterilized, have a negative dipstick testing or a negative serum testing or patients who are postmenopausal) 4. Characteristics of the treatment We will be using ropivacaine - naropin 7,5mg/ml, a local anaesthetic of the amide type. The administered dose of this local anaesthetic will be 3mg/kg for each patient. Depending on the study group the patient belongs to, this dose will be given in full by either local injection at the trocar entry points or by intraperitoneal injection or it will be divided between both injection sites, respectively 1mg at the trocar sites and 2mg intraperitoneal. The unequal dose distribution is based on the surface area the local anaesthetic has to cover.

5. Methodology Anaesthetic management will be standardized for each person. The anaesthetist will insert an intravenous line and connect the patient to the monitor. We will be using routine intraoperative monitoring devices such as an electrocardiograph, a pulse oximetry and a non-invasive blood pressure monitor. The patient is preoxygenated with 100% O2 before induction.

Anaesthetic protocol

Induction:

* fentanyl 2μg/kg
* Propofol TCI marsh model 6μg/ml - titration based on effect
* Rocuronium 0.5mg/kg

Maintenance:

- Propofol TCI Marsh model: 4μ/ml - (8-12mg/kg/u) - titration based on effect, blood pressure and heart rate.

Analgesia intraoperatively:

* Ketorolac 30mg at induction (if no contraindications; and > 60kg; if the patient weight is < 60kg the dose will be lowered to 20mg)
* Paracetamol 1g one half hour before the end of the surgery Different study groups

At the end of the successful gynaecologic laparoscopy, patients will receive the additional pain management according to their randomly assigned study group:

* Group A patients will receive 1) intra-abdominal instillation 0.75% Ropivacaine 2 mg / kg in 200 ml of NaCl through the trocars and 2) Infiltration of the surgical wounds at the trocar sites with 0.75% Ropivacaine 1 mg / kg in 20 ml of NaCl (Sodiumchloride)
* Group B patients will receive infiltration of the surgical wounds at the trocar sites with 0.75% Ropivacaine 3 mg / kg in 20 ml of NaCl.
* Group C patients will receive intra-abdominal instillation 0.75% Ropivacaine 3 mg / kg in 200 ml of NaCl through the trocars.

Suction and aspiration is avoided after instillation of local anaesthetic intra-abdominal in group A and C.

The study medication will be prepared in the operating room right before use. This means that neither the anaesthesiologist nor the surgeon, performing the surgery, are blinded. This isn't a problem since it is already at the end of the procedure and they will not be the ones following up on the patients for study purposes.

End of the procedure After surgery, the patients will be transferred to the recovery room. A standard postoperative analgesic regimen will be used in all patients with Numeric Rating Scale (NRS) >= 3.

As long as the patient is in the hospital, she will receive paracetamol 1g every 6 hours, preferably given orally. If, despite this regimen, the NRS score is higher than 3, they will receive tramadol 100mg IV + alizapride 50 mg. There will be a re-evaluation after 30 minutes. If the NRS is still higher than 3, an anaesthesiologist will be consulted and a subcutaneous dose of morphine will be given. The dose will be 5 mg if the body weight of the patient is less than 90 kg and the patient is less than 70 years old. In a patient heavier than 90 kg and younger than 70 years, the dose will be 10mg morphine subcutaneously.

The nurses of the day hospital will complete the first page(s) of the patient's questionnaire.

Later that day the patient will be discharged from the hospital if all the discharge criteria are met according to standard operating procedures.

When going home all patients receive a map with their questionnaire, a prescription for paracetamol 1g if necessary, max 4 times a day, and a last reminder to not forget about the questionnaire. In this study, we will focus about the first week postoperatively.

6. Questionnaire In total 7 parameters will be questioned: abdominal pain, shoulder pain, nausea, vomiting, itching, urinating and activity level. The questionnaire that will be given to the patients consists of an introduction page and 5 identical questionnaires. Assessment will take place at respectively 1 h, 2 h, 6 h, 24 h and 1 w postoperatively. Abdominal pain will be scored by the patients using the numeric rating scale. The patients will be asked to rate the severity of pain via NRS ranging from no pain (score 0) to the worst possible pain (score 10).

This method is explained in the introduction page and is the method of choice to evaluate pain in the recovery room. This means that all the patients will already be familiar with the scoring system before going home. Intra-abdominal pain will be assessed during rest and during an effort, for example coughing. In the postoperative period, the time to first analgesic administration and total analgesic requirements (paracetamol, tramadol and morphine) will be recorded.

For the other parameters, our interests lie in the presence or absence of these elements so we chose for a simple "yes" or "no" question.

The individuals filling in the questionnaires, the patients or the nurses of the recovery room will always be blinded to the study groups, as will the nurse contacting the patients for the follow up. The research nurses will contact the patients through telephone 24 h after surgery and again 1 week after surgery to get the answers of the questionnaires. They will be unaware of the study group the patient was subdivided into. The responses will be recorded and analysed by members of the research group. If the patients are not pain free after one week, we will contact them again after one month. After that, they will be called once a month until they are pain free or 6 months have passed. Postoperative pain lasting more than one week could be and indicator for the onset of chronic pain. (13) However, this topic will need additional research that, for the moment, is beyond the scope of our investigation.

7. Statistics: Comparison of the categorical or ordinal variables will be performed using Chi square or Fisher exact test and relative risk with 95 % confidence intervals as appropriate Continuous variables will be presented in median values and will be compared using ANOVA. Multivariate logistic regression analysis will be performed. P values of less than 0.05 will be regarded statistically significant. All the calculations will be performed with the SPSS 11.0 statistical package (SPSS, Inc., Chicago, IL) (Dupont WD, Plummer WD, http://www.spss.com). According to that the sample size should be at least 16 cases for each group when we want the power of the study to be 80%.æ

ELIGIBILITY:
Inclusion Criteria:

1. Elective gynecologic laparoscopy for benign conditions at Antwerp University Hospital.
2. Successful laparoscopy without surgical or anesthetic complications.
3. Female
4. 18-70 years
5. ASA I-II

Exclusion Criteria:

1. Hypersensitivity to anaesthetics of the amide-type
2. Obesity, BMI > 35
3. Patients with chronic use of analgesics / chronic pain
4. Patients with an abnormal liver function
5. Urgent surgical procedures
6. Pregnancy (this means we only include patients who use contraceptives, are sterilized, have a negative dipstick testing or a negative serum testing or patients who are postmenopausal)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Abdominale Pain scores postoperatively | one week
  Numeric rating scale NRS
need of pain medication postoperatively | one week
  note in file

SECONDARY OUTCOMES:
postoperative nausea and vomiting | one week
  score yes/no
shoulder pain postoperatively | one week
  score yes/no
itching postoperatively | one week
  score yes/no
problems with urinating postoperatively | one week
  score yes/no
Activity level postoperatively: return to normal | one week
  score yes/no

CONTACTS AND LOCATIONS:
Locations (1):
- UZA, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided